CLINICAL TRIAL: NCT01287949
Title: An Open-label, Multicentre Study to Evaluate the Immunogenicity and Safety of One Dose of a Diphtheria, Tetanus, Acellular Pertussis and Poliomyelitis Vaccine (REPEVAX) Followed by 2 Doses of a Diphtheria, Tetanus and Poliomyelitis Vaccine (REVAXIS) in Subjects of 40 Years of Age or Older Without a Previous Diphtheria- and Tetanus-containing Booster Within the Last 20 Years
Brief Title: Safety and Immunogenicity Study of a Diphtheria, Tetanus, Acellular Pertussis and Poliomyelitis Vaccine (REPEVAX) Followed by 2 Doses of a Diphtheria, Tetanus and Poliomyelitis Vaccine (REVAXIS) in Subjects of 40 Years of Age or Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RPV04C
Record Dates: First submitted 2011-01-31; First posted 2011-02-02 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Diphtheria; Tetanus; Poliomyelitis; Pertussis
Keywords: Diphtheria; Tetanus; Poliomyelitis; Pertussis (acellular); Biological/vaccine
MeSH Terms: conditions — Diphtheria; Tetanus; Poliomyelitis; Whooping Cough | interventions — Tetanus Toxoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- REPEVAX followed by REVAXIS administration (Experimental)
  Interventions: Biological: Diphtheria, tetanus, polio and pertussis vaccination

INTERVENTIONS:
Biological: Diphtheria, tetanus, polio and pertussis vaccination — 1 dose of REPEVAX (0.5 mL) at Day 0, 1 dose of REVAXIS (0.5 mL) 1 month later and 1 dose of REVAXIS 6 month later

SUMMARY:
Primary objective:

* To demonstrate that 3 doses of a vaccine containing Td-IPV valences administered in a 0, 1 and 6-month schedule induce an acceptable immune response in terms of seroprotection rates (SPR) against diphtheria, tetanus and poliomyelitis 1, 2 and 3, in subjects of 40 years of age or older with no diphtheria- and tetanus-containing booster within the last 20 years
* To evaluate the percentage of subjects with antibody titre ≥5 EU/mL (ELISA) for each of the pertussis components (PT, FHA, PRN and FIM) after 1 dose of REPEVAX in these subjects

Secondary objectives:

* If the primary objective is achieved, to determine whether 1 or 2 doses of a vaccine containing Td-IPV valences induce an acceptable response in terms of seroprotection rates (SPR) against diphtheria, tetanus and poliomyelitis 1, 2 and 3, in subjects of 40 years of age or older with no diphtheria- and tetanus-containing booster within the last 20 years
* To describe the immune responses to REPEVAX in these subjects
* To describe the immune responses to REVAXIS administered 1 and 6 months after the administration of REPEVAX in these subjects

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥40 years
* No receipt of a booster dose with a tetanus-, diphtheria-containing vaccine within the last 20 years

Exclusion Criteria:

* Medically diagnosed pertussis disease within the last 10 years
* Receipt of medication / vaccine that may interfere with study assessments
* Febrile illness or moderate or severe acute illness/infection
* Know pregnancy
* History of hypersensitivity or anaphylactic or other allergic reactions to any of the vaccine components, or history of a life-threatening reaction to the study vaccines or a vaccine containing any of the same substances
* History of Guillain Barré syndrome or brachial neuritis following a previous vaccination
* History of encephalopathy of unknown origin within 7 days after immunization with a pertussis-containing vaccine or neurological disorders
* Known or suspected immune dysfunction
* Thrombocytopenia, bleeding disorder or anticoagulants contraindicating intramuscular vaccination
* Chronic disease or intercurrent illness that might interfere with study assessments

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Diphtheria seroprotection rate | 28 to 35 days afeter each vaccine administration
Tetanus seroprotection rate | 28 to 35 days after each vaccine administration
Polio seroprotection rate | 28 to 35 days after each vaccine administration
Pertussis response rate | 28 to 35 days after REPEVAX administration

SECONDARY OUTCOMES:
Solicited injection-site reactions, solicited systemic reactions | From day 0 to day 7 following REPEVAX and REVAXIS vaccination
Unsolicited injection-site adverse reactions and systemic adverse events | From day 0 to day 28 following REPEVAX and REVAXIS vaccination
Number and proportion of Serious adverse events | From the first vaccination to the last visit of the subject

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (12):
- France (6):
  - Sanofi Pasteur MSD investigational site, Clermont-Ferrand
  - Sanofi Pasteur MSD investigational site, Lille
  - Sanofi Pasteur MSD investigational site, Montpellier
  - Sanofi Pasteur MSD investigational site, Paris
  - Sanofi Pasteur MSD investigational site, Poitiers
  - Sanofi Pasteur MSD investigational site, Saint-Etienne
- Germany (6):
  - Sanofi Pasteur MSD investigational site, Balve
  - Sanofi Pasteur MSD investigational site, Berlin
  - Sanofi Pasteur MSD investigational site, Dülmen
  - Sanofi Pasteur MSD investigational site, Nuremberg
  - Sanofi Pasteur MSD investigational site, Offenbach
  - Sanofi Pasteur MSD investigational site, Rodgau